CLINICAL TRIAL: NCT06964724
Title: NeVa International, MulTi-center, Retrospective cOmparative Stent Retriever Study
Brief Title: NeVa Retrospective Comparative SR Study
Acronym: NITRO
Status: Active, not recruiting | Type: Observational
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Other Study IDs: VS-010
Record Dates: First submitted 2025-04-18; First posted 2025-05-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stroke Acute
Keywords: NeVa; Mechanical Thrombectomy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients experiencing acute ischemic stroke due to large vessel occlusion: According to Guidelines AIS patients due to LVO should receive mechanical thrombectomy (with a stent retriever) under certain conditions.
  Interventions: Procedure: Mechanical thrombectomy

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Mechanical thrombectomy with stent retriever

SUMMARY:
To compare safety and effectiveness of NeVa Stent Retriever (SR) to Control SR in the treatment of stroke caused by large vessel occlusion. The main questions it aims to answer are:

How do recanalization rates for NeVa SR compare with those of the Control SR? How does NeVa SR safety compare with Control SR safety?

DETAILED DESCRIPTION:
NITRO is a multicenter, retrospective, comparative, non-inferiority, cohort study designed to compare NeVa SR with Control SR for safety and effectiveness when removing thrombus in subjects presenting with acute ischemic stroke (AIS) due to large vessel occlusion (LVO). The objective of the NeVa International, Multi-center, Retrospective Comparative stent retriever (SR) study (NITRO) study is to compare safety and effectiveness of the NeVa SR to commonly used SR with CE-mark, and US FDA clearance, to restore blood flow in patients experiencing acute ischemic stroke due to large intracranial vessel occlusion. NITRO aims to collect data describing real-world clinical practices when using SRs according to their indicated use within the indicated population. As such, the eligibility criteria define patients who are diagnosed with AIS and are indicated for endovascular MT aligning to the target population for the proposed device. The present study will include data from subjects treated with either NeVa SR or one of the Control SR. Control SR will include any SR commonly used in thrombectomy trials as first-line strategies and which represent CE-mark, and US FDA cleared stent retrievers.

ELIGIBILITY:
Inclusion Criteria:

* Treatment during the enrollment period
* Age ≥18
* Baseline modified Thrombolysis in Cerebral Infarction (mTICI) score ≤ 1
* Pre-stroke modified Rankin score (mRS) of 0 or 1
* Internal Carotid Artery (ICA), Middle Cerebral Artery (first segment M1/ second segment M2), basilar artery or vertebral artery occlusion
* National Institutes of Health Stroke Scale (NIHSS) score ≥ 8 and ≤ 25
* Thrombectomy procedure initiated within 8h of Time Last Known Well (TLKW)
* Intravenous Tissue Plasminogen Activator (IV-tPA) failed, given within 3h of TLKW, or ineligibility for thrombolytic drug

Exclusion Criteria:

* First line contact aspiration alone or non-study device as first-line device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from acute ischemic stroke from large vessel occlusion treated with study device.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Reperfusion Effectiveness | Procedural
  Number of patients with a Modified Thrombolysis in cerebral infarction (mTICI) ≥2B and mTICI≥2C recanalization after 1st pass and at end of procedure

SECONDARY OUTCOMES:
Procedural symptomatic bleeding events | Within 24 hours post intervention
  Number of patients experiencing symptomatic intracranial hemorrhage (sICH)
Procedure Safety | Within 24 hours post intervention
  Number of patients experiencing procedure related serious Adverse Events (PRSAE)
Device relationship to serious adverse events | Within 24 hours post intervention
  Number of patients experiencing a serious adverse device effect (SADE)

OTHER OUTCOMES:
Functional Independence at 90 days | At 90 Days
  Number of patients with a Modified Rankin Scale (mRS) 0-2
90-day Mortality | Within 90 days post intervention
  Number of patients that died at 90-days from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuijpers, MSc, Study Director — Vesalio
Locations (5):
- Hospital Espanol de Mendoza, Mendoza, Argentina
- CHU LIege, Liège, Belgium
- UK Munster, Münster, Germany
- Republican Vilnius University Hospital, Vilnius, Lithuania
- İstanbul Aydrn Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this stage not yet discussed how or at which URL the Protocol defined Endpoints will be made available.